CLINICAL TRIAL: NCT00049543
Title: A Phase III Prospective Randomized, Double-Blind, Placebo-Controlled Trial of the Epidermal Growth Factor Receptor Antagonist, ZD1839 (IRESSA) in Completely Resected Primary Stage IB, II and IIIA Non-Small Cell Lung Cancer
Brief Title: Gefitinib in Treating Patients With Stage IB, II, or IIIA Non-small Cell Lung Cancer That Was Completely Removed by Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2014-00650; NCI-2014-00650 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SWOG-CAN-NCIC-BR19; ECOG-CAN-NCIC-BR19; BR19; CDR0000258118; CAN-NCIC-BR19; BR.19 (Other: National Cancer Institute of Canada Clinical Trials Group); BR.19 (Other: CTEP); NCT00953069 (obsolete NCT alias)
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Results first posted 2015-01-01 (Estimated); Last update posted 2015-01-01 (Estimated); Status verified 2014-03

CONDITIONS: Adenocarcinoma of the Lung; Adenosquamous Cell Lung Cancer; Bronchoalveolar Cell Lung Cancer; Large Cell Lung Cancer; Squamous Cell Lung Cancer; Stage IB Non-small Cell Lung Cancer; Stage IIA Non-small Cell Lung Cancer; Stage IIB Non-small Cell Lung Cancer; Stage IIIA Non-small Cell Lung Cancer
MeSH Terms: conditions — Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar; Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (gefitinib) (Experimental): Patients receive gefitinib PO QD for 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: gefitinib; Other: laboratory biomarker analysis
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO QD for 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: placebo; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: gefitinib — Given PO
  Other Names: Iressa; ZD 1839
  Arms: Arm I (gefitinib)
Other: placebo — Given PO
  Other Names: PLCB
  Arms: Arm II (placebo)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase III trial studies how well gefitinib works in treating patients with stage IB, II, or IIIA non-small cell lung cancer that was completely removed by surgery. Gefitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known if gefitinib may be an effective treatment in preventing tumors from returning after they have been removed by surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess, in comparison with placebo, the impact of adjuvant therapy with two years of daily oral ZD1839 (IRESSA) (gefitinib) on the overall survival of patients with completely resected (T1N1-2, T2N0-2, T3N0-2) non-small cell lung cancer (NSCLC).

SECONDARY OBJECTIVES:

I. To compare the disease-free survival in the placebo arm to the ZD1839 (IRESSA) arm.

II. To confirm the prognostic significance of epidermal growth factor receptor (EGFR) expression, phosphorylation and mutations when present in the primary tumor.

III. To assess the ability of EGFR expression, phosphorylation and mutations in the primary tumor to predict the relative impact of ZD1839 (IRESSA) on survival.

IV. To establish a comprehensive tumour bank linked to a clinical database for the further study of molecular markers in resected NSCLC.

V. To further evaluate toxicity related to ZD1839 (IRESSA).

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive gefitinib orally (PO) once daily (QD) for 2 years in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive placebo PO QD for 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 6 months, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histological proof of a primary non-small cell lung cancer (bronchoalveolar carcinomas presenting as a discrete solitary radiological mass or nodule are eligible)
* Patients must be classified post-operatively as stage IB, II or IIIA on the basis of pathologic criteria
* At the time of resection a complete mediastinal lymph node resection or at least lymph node sampling should have been attempted; if a complete mediastinal lymph node resection or lymph node sampling was not undertaken, any mediastinal lymph node which measured 1.5 cm or more on the pre-surgical computed tomography (CT)/magnetic resonance imaging (MRI) scan or any area of increased uptake in the mediastinum on a pre-surgical positron emission tomography (PET) scan must have been biopsied; note: a pre-surgical PET scan is not mandatory

  * The nodal tissue must be labelled according to the recommendations of the American Thoracic Society; surgeons are encouraged to dissect or sample all accessible nodal levels; the desirable levels for biopsy are:

    * Right upper lobe: 4, 7, 10
    * Right middle lobe: 4, 7, 10
    * Right lower lobe: 4, 7, 9, 10
    * Left upper lobe: 5, 6, 7, 10
    * Left lower lobe: 7, 9, 10
* Surgery may consist of lobectomy, sleeve resection, bilobectomy or pneumonectomy as determined by the attending surgeon based on the intraoperative findings; patients who have had only segmentectomies or wedge resections are not eligible for this study; all gross disease must have been removed at the end of surgery; all surgical margins of resection must be negative for tumor
* No more than 16 weeks may have elapsed between surgery and randomization; for patients who received post-operative adjuvant platinum-based chemotherapy, no more than 26 weeks may have elapsed between surgery and randomization
* Patient must consent to provision of and investigator(s) must agree to submit a representative formalin fixed paraffin block of tumor tissue at the request of the Central Tumor Bank in order that the specific EGFR correlative marker assays may be conducted
* The patient must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Leukocytes >= 3.0 x 10^9/L or >= 3000/ul
* Absolute granulocyte count >= 1.5 x 10^9/L or >= 1,500/ul
* Platelets >= 100 x 10^9/L or >= 100,000/ul
* Total bilirubin within normal institutional limits
* Alkaline phosphatase =< 2.5 x institutional upper limit of normal; if alkaline phosphatase is greater than the institutional upper limit of normal (UNL) but less than the maximum allowed, an abdominal (including liver) ultrasound, CT or MRI scan and a radionuclide bone scan must be performed prior to randomization to rule out metastatic disease; if the values are greater than the maximum allowed, patients will not be considered eligible regardless of findings on any supplementary imaging
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and/or alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal; if AST (SGOT) or ALT (SGPT) are greater than the institutional upper limit of normal (UNL) but less than the maximum allowed, an abdominal (including liver) ultrasound, CT or MRI scan must be performed prior to randomization to rule out metastatic disease; if the values are greater than the maximum allowed, patients will not be considered eligible regardless of findings on any supplementary imaging
* Patient must have a chest x-ray done within 14 days prior to randomization; patient must have a CT or MRI scan of the chest done within 90 days prior to surgical resection if at least one of the following was undertaken:

  * A complete mediastinal lymph node resection; or
  * Biopsy of all desired levels of lymph nodes - as specified above; or
  * A pre-surgical PET scan within 60 days prior to surgical resection If none of the above was undertaken then the CT or MRI scan of the chest must have been performed within 60 days prior to surgical resection Note: a pre-surgical PET scan is not mandatory
* Patient must have an electrocardiogram (EKG) done within 14 days prior to randomization
* Women of childbearing age and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and while taking study medication and for a period of three months after final dose; should a woman become pregnant or suspect she is pregnant while she or her male partner are participating in this study, she should inform her treating physician immediately
* Patients may receive post-operative radiation therapy; patients must have completed radiation at least 3 weeks prior to randomization and have recovered from all radiation-induced toxicity; patients who have received radiation therapy should also be randomized within 16 weeks of surgery
* Patient consent must be obtained according to local institutional and/or University Human Experimentation Committee requirements; it will be the responsibility of the local participating investigators to obtain the necessary local clearance, and to indicate in writing to either the National Cancer Institute of Canada (NCIC) Clinical Trials Group (CTG) study coordinator (for NCIC CTG centers) or the Cancer Trials Support Unit (CTSU) (for all other investigators), that such clearance has been obtained, before the trial can commence in that center; a standard consent form for the trial will not be provided, but a sample form is given; this sample consent form has been approved by the National Cancer Institute (NCI) Central Institutional Review Board (IRB) and must be used unaltered by those CTSI centers which operate under CIRB authority; for NCIC CTG centers, a copy of the initial full board Research Ethics Board (REB) approval and approved consent form must be sent to the NCIC CTG central office; please note that the consent form for this study must contain a statement which gives permission for the government agencies, NCI, NCIC CTG and monitoring agencies to review patient records

  * NCIC-CTG Centers: the patient must have the ability to understand and the willingness to sign a written informed consent document; the patient must sign the consent form prior to randomization
  * CTSU Centers: the patient, or in the case of a mentally incompetent patient his or her legally authorized and qualified representative, must have the ability to understand and the willingness to sign a written informed consent document; the consent form must be signed prior to randomization
* Patients must be accessible for treatment and follow-up; investigators must assure themselves that patients registered on this trial will be available for complete documentation of the treatment administered, toxicity and follow-up
* Initiation of protocol treatment must begin within 10 working days of patient randomization
* Patients may have received post-operative adjuvant platinum-based chemotherapy; patients must have completed chemotherapy at least 3 weeks prior to randomization and have recovered from all chemotherapy-induced toxicity; patients who have received adjuvant chemotherapy should also be randomized within 26 weeks of surgery

Exclusion Criteria:

* Prior or concurrent malignancies; patients who have had a previous diagnosis of cancer, if they remain free of recurrence and metastases five years or more following the end of treatment and, in the opinion of the treating physician do not have a substantial risk of recurrence of the prior malignancy, are eligible for the study; patients who have been adequately treated for non-melanomatous skin cancer or carcinoma in situ of the cervix are eligible irrespective of when that treatment was given
* A combination of small cell and non-small cell carcinomas or a pulmonary carcinoid tumor
* More than one discrete area of apparent primary cancer (even if within the same lobe, T4, IIIB)
* Clinically significant or untreated ophthalmologic (e.g. Sjogren's etc.) or gastrointestinal conditions (e.g. Crohn's disease, ulcerative colitis)
* Any active pathological condition that would render the protocol treatment dangerous such as: uncontrolled congestive heart failure, angina, or arrhythmias, active uncontrolled infection, or others
* A history of psychiatric or neurological disorder that would make the obtainment of informed consent problematic or that would limit compliance with study requirements
* Patient, if female, is pregnant or breast-feeding
* Neoadjuvant chemotherapy or immunotherapy for NSCLC; however, patients may have received pre-operative limited field, low dose (less than 1000 cGy) external beam radiation therapy or endobronchial brachytherapy or laser therapy for short term control of hemoptysis or lobar obstruction; full dose pre-operative radiotherapy of curative intent is a cause for exclusion; patients may have received post-operative adjuvant platinum-based chemotherapy however non-platinum-based chemotherapy is a cause for exclusion
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the agents used on this trial; patients with ongoing use of phenytoin, carbamazepine, barbiturates, rifampicin, or St John's Wort are excluded
* Incomplete healing from previous oncologic or other major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2002-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glennwood Goss, Principal Investigator — Canadian Cancer Trials Group
Locations (1):
- National Cancer Institute of Canada Clinical Trials Group, Kingston, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Gefitinib) | Arm II (Placebo)
Started | 251 | 252
Completed | 249 | 243
Not Completed | 2 | 9
Not completed — still on treatment | 2 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Gefitinib) | Arm II (Placebo) | Total
Number analyzed (Participants) | 251 | 252 | 503
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 105 | 120 | 225
  >=65 years | 146 | 132 | 278
Age, Continuous [Median (Full Range); unit: years] | 67.3 [38.9 to 88] | 65.9 [30.4 to 86.9] | 66.7 [30.4 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 116 | 232
  Male | 135 | 136 | 271
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 6 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 10 | 9 | 19
  White | 233 | 235 | 468
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 52 | 50 | 102
  United States | 199 | 202 | 401

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: The survival experience of patients in both treatment groups will be described by the Kaplan-Meier method. A stratified log-rank test will be used as the primary method to compare the overall survival between two arms adjusting for the stratification factors. An unadjusted analysis will also be performed. Five years survival rate will be reported.
Time Frame: From randomization to the time of death from any cause, assessed up to 5 years
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of 5 years survival rate
Arm/Group | Arm I (Gefitinib) | Arm II (Placebo)
Number analyzed (Participants) | 251 | 252
percentage of 5 years survival rate | 0.52 [0.44 to 0.58] | 0.57 [0.51 to 0.64]
Statistical Analysis 1: Comparison: Arm I (Gefitinib) vs Arm II (Placebo); The Kaplan-Meier estimates of survival distribution for overall survival by treatment arm are reported, and the log rank test stratified by the stratification factors at randomization (exclude center) was used to compare the difference in the overall survival between two treatment arms. Hazard ratio of comparison of study treatment arm to placebo and it 95% C.I. were reported; Test type: Superiority or Other; p = 0.14, Log Rank; Hazard Ratio (HR) = 1.24, 95% CI 2-sided [0.94 to 1.64]

2. Secondary Outcome: Disease Free Survival
Description: The survival experience of patients in both treatment groups will be described by the Kaplan-Meier method. A stratified log-rank test will be used as the primary method to compare the disease free survival between two arms adjusting for the stratification factors. Five years disease free survival rate will be reported.
Time Frame: From randomization to the time of documented recurrence of the primary cancer, assessed up to 5 years
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of 5-year disease free rate
Arm/Group | Arm I (Gefitinib) | Arm II (Placebo)
Number analyzed (Participants) | 251 | 252
percentage of 5-year disease free rate | 0.49 [0.42 to 0.55] | 0.56 [0.50 to 0.63]
Statistical Analysis 1: Comparison: Arm I (Gefitinib) vs Arm II (Placebo); Test type: Superiority or Other; p = 0.15, Log Rank — Stratified by stratification factors at randomization (except center); Stratified by stratification factors at randomization (except center); Hazard Ratio (HR) = 1.22, 95% CI 2-sided [0.93 to 1.61]

3. Secondary Outcome: Incidence of Toxicities Graded Using the NCI Common Terminology Criteria for Adverse Events Version 3.0
Description: The incidence of toxicities will be summarized by type of adverse event and severity. A Fisher's exact test will be used to compare toxicities between the two arms.
Time Frame: Up to 5 years
Population: All patients who received at least 1 dose of the treatment
Measure: Number; unit: participants
Arm/Group | Arm I (Gefitinib) | Arm II (Placebo)
Number analyzed (Participants) | 249 | 243
participants | 229 | 153

ADVERSE EVENTS:
Arm/Group | Arm I (Gefitinib) | Arm II (Placebo)
Serious Adverse Events (participants affected / at risk) | 34/249 | 43/243
Other Adverse Events (participants affected / at risk) | 240/249 | 226/243
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Gefitinib) (N=249) | Arm II (Placebo) (N=243)
Cardiac General - Other (Cardiac disorders) | 2 | 4
Cardiac ischemia/infarction (Cardiac disorders) | 1 | 1
Left ventricular diastolic dysfunction (Cardiac disorders) | 1 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 0
Blurred vision (Eye disorders) | 1 | 0
Ocular - Other (Eye disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 4 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0
Fistula, GI Small bowel NOS (Gastrointestinal disorders) | 0 | 1
GI - Other (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Heartburn (Gastrointestinal disorders) | 1 | 1
Hemorrhage, GI Colon (Gastrointestinal disorders) | 1 | 0
Hemorrhage, GI Lower GI NOS (Gastrointestinal disorders) | 1 | 0
Hemorrhage, GI Upper GI NOS (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Pain Abdomen NOS (Gastrointestinal disorders) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Constitutional Symptoms - Other (General disorders) | 0 | 2
Death Disease progression NOS (General disorders) | 1 | 0
Edema: limb (General disorders) | 0 | 2
Fatigue (General disorders) | 2 | 1
Fever (General disorders) | 2 | 1
Pain - Other (General disorders) | 1 | 0
Pain Chest/thorax NOS (General disorders) | 0 | 4
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Liver dysfunction (Hepatobiliary disorders) | 2 | 0
Allergic reaction (Immune system disorders) | 0 | 1
Infection - Other (Infections and infestations) | 4 | 3
Infection with normal ANC Lung (Infections and infestations) | 1 | 1
Infection with unknown ANC Lung (Infections and infestations) | 0 | 2
Fracture (Injury, poisoning and procedural complications) | 2 | 0
ALT (Investigations) | 0 | 1
AST (Investigations) | 0 | 1
Creatinine (Investigations) | 0 | 1
Weight gain (Investigations) | 1 | 0
Weight loss (Investigations) | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain Bone (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain Extremity-limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain Joint (Musculoskeletal and connective tissue disorders) | 1 | 1
Ataxia (Nervous system disorders) | 1 | 0
CNS hemorrhage (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Neuropathy-sensory (Nervous system disorders) | 1 | 1
Pain Head/headache (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Speech impairment (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 2
Mood alteration Anxiety (Psychiatric disorders) | 2 | 2
Mood alteration Depression (Psychiatric disorders) | 0 | 1
Psychosis (Psychiatric disorders) | 0 | 1
Renal - Other (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 1 | 1
ARDS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 | 14
Fistula, pulmonary Lung (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hemorrhage pulmonary Lung (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hemorrhage pulmonary Respiratory tract NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pain Pleura (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Hand-foot (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 1
Peripheral arterial ischemia (Vascular disorders) | 0 | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 4 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Gefitinib) (N=249) | Arm II (Placebo) (N=243)
Constipation (Gastrointestinal disorders) | 39 | 33
Diarrhea (Gastrointestinal disorders) | 155 | 75
Heartburn (Gastrointestinal disorders) | 19 | 20
Nausea (Gastrointestinal disorders) | 66 | 45
Pain Abdomen NOS (Gastrointestinal disorders) | 18 | 7
Vomiting (Gastrointestinal disorders) | 32 | 19
Edema: limb (General disorders) | 11 | 14
Fatigue (General disorders) | 135 | 130
Pain Chest/thorax NOS (General disorders) | 86 | 107
Infection - Other (Infections and infestations) | 19 | 20
ALT (Investigations) | 13 | 3
AST (Investigations) | 14 | 2
Weight loss (Investigations) | 16 | 6
Anorexia (Metabolism and nutrition disorders) | 70 | 40
Hyperglycemia (Metabolism and nutrition disorders) | 26 | 23
Pain Back (Musculoskeletal and connective tissue disorders) | 13 | 17
Pain Bone (Musculoskeletal and connective tissue disorders) | 11 | 15
Pain Joint (Musculoskeletal and connective tissue disorders) | 14 | 23
Pain Muscle (Musculoskeletal and connective tissue disorders) | 12 | 23
Dizziness (Nervous system disorders) | 17 | 17
Neuropathy-sensory (Nervous system disorders) | 26 | 38
Pain Head/headache (Nervous system disorders) | 19 | 15
Insomnia (Psychiatric disorders) | 12 | 19
Mood alteration Anxiety (Psychiatric disorders) | 16 | 11
Mood alteration Depression (Psychiatric disorders) | 14 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 63 | 71
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 130 | 147
Hemorrhage pulmonary Nose (Respiratory, thoracic and mediastinal disorders) | 16 | 4
Acne (Skin and subcutaneous tissue disorders) | 13 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 22 | 14
Dry skin (Skin and subcutaneous tissue disorders) | 107 | 46
Nail changes (Skin and subcutaneous tissue disorders) | 13 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 92 | 32
Rash (Skin and subcutaneous tissue disorders) | 167 | 66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less